CLINICAL TRIAL: NCT05030883
Title: The Effect of Source Type and Protective Message on the Critical Evaluation of News Messages on Facebook: An Experimental Study in the Netherlands.
Brief Title: The Effect of a Protective Message on Critical Evaluation of Fake News
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Responsible Party: Principal Investigator, Frans Folkvord, Assistant professor, Tilburg University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TiU-1
Record Dates: First submitted 2021-08-03; First posted 2021-09-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2021-08

CONDITIONS: Disclosure of Protective Message

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- unreliable source (Experimental): In this condition participants receive a news message from an unreliable source
  Interventions: Behavioral: Source of news
- reliable source (Experimental): In this condition participants receive a news message from an reliable source
  Interventions: Behavioral: Source of news
- no source (Experimental): In this condition participants receive a news message without a source
  Interventions: Behavioral: Source of news

INTERVENTIONS:
Behavioral: Source of news — The main intervention was the source of the news that was shown to participants

SUMMARY:
Background: Disinformation has become an increasing societal concern, especially due to the speed that news is shared in the current digital era. In particular in the healthcare sector disinformation can lead to serious casualties, as the current COVID-19 crisis clearly shows.

Objective: The main aim of this study was to experimentally examine the effects of information about the source's and a displayed protective warning message on users' critical evaluation of news items, as well as the perception of accuracy of the news item.

Methods: A 3(unreliable versus reliable versus no identified source) x 2 (protective message: with versus without) between subject design has been conducted among 307 participants (mean age = 29 years, SD = 10.9 years).

ELIGIBILITY:
Inclusion Criteria:

* Facebook user
* older than 18
* Dutch

Exclusion Criteria:

* younger than 18 years
* no facebook

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Critical evaluation of source and news | immediately after exposure, 5 minutes
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tilburg School of Humanities and Digital Sciences, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request we will decide to share the data with other researchers

REFERENCES:
- [Derived] Folkvord F, Snelting F, Anschutz D, Hartmann T, Theben A, Gunderson L, Vermeulen I, Lupianez-Villanueva F. Effect of Source Type and Protective Message on the Critical Evaluation of News Messages on Facebook: Randomized Controlled Trial in the Netherlands. J Med Internet Res. 2022 Mar 31;24(3):e27945. doi: 10.2196/27945. PMID 35357314